CLINICAL TRIAL: NCT04221464
Title: Development of a Clinical and Biological Database Monocentric and Prospective in Peritoneal Carcinosis
Brief Title: Development of a Clinical and Biological Database in Peritoneal Carcinosis (BCB CARCINOSE)
Acronym: BCB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2019-01 BCA
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Peritoneal Carcinosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumors and blood collection (Experimental): For all the patients include in the study :
  * Blood samples will be collected at different times : before any treatment, at every surgery, one month after any surgery, at progression.
  * Tumours and not tumours tissues will be collected at different times : Before any surgery, one month after any surgery
  In parallel to this biological collection, standardized clinical data will be entered into a database treatment, at every surgery
  Interventions: Biological: biological collection; Other: Tissues collections

INTERVENTIONS:
Biological: biological collection — Blood samples collected before any treatment (if chemotherapy for example), at every surgery, one month after surgery, at progression
Other: Tissues collections — Tumours and not tumours tissues will be collected before any treatment (if chemotherapy for example), at every surgery, one month after surgery, at progression

SUMMARY:
The creation of a prospective clinical-biological base dedicated to peritoneal carcinosis must therefore be able to serve as a support for this essential search for transfer.

DETAILED DESCRIPTION:
The main objective is to improve the knowledge of carcinosis mechanisms to develop a specific treatment.

That's why this blood collection and tissue collection is very important for the future, these collection will be permitted to the scientists to develop a research specially for carcinosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18;
* Patient managed for peritoneal carcinosis : digestives origins (pancreatic, gastroesophageal junction, colorectal, bowel) or peritoneum cancer
* Patient eligible for a peritoneal carcinosis treatment : at least one (or more) surgery (s) ;chemotherapy or any treatment for this disease
* Patient agree will all study procedure : biological samples & tissues samples
* Patient giving informed consent

Exclusion Criteria:

* Patient not affiliated to Social Protection system
* Patient unable to understand or comply with study instructions or requirements for psychological, family, social or geographical reasons
* The level of French is insufficient to consent to the study and to response to the questionnaires
* Patient under guardianship
* Pregnancy ou breast-feeding women
* Patient treated in case of an emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2038-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who gave their consent to participate in the study | Until the study completion: 4 years
  The proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Overall Officials: François QUENET,MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- Institut du cancer de Montpellier ICM, Montpellier, France